CLINICAL TRIAL: NCT00014235
Title: Nonmyeloablative PBSC Allografting From HLA Matched Related Donors Using Fludarabine and/or Low Dose TBI With Disease-Risk Based Immunosuppression
Brief Title: Fludarabine Phosphate and Total-Body Radiation Followed by Donor Peripheral Blood Stem Cell Transplant and Immunosuppression in Treating Patients With Hematologic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1596.00; NCI-2012-00671 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1596.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Acute Myeloid Leukemia/Transient Myeloproliferative Disorder; Acute Undifferentiated Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Blastic Plasmacytoid Dendritic Cell Neoplasm; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Burkitt Lymphoma; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Myelomonocytic Leukemia; Cutaneous B-cell Non-Hodgkin Lymphoma; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Juvenile Myelomonocytic Leukemia; Mast Cell Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Primary Systemic Amyloidosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage II Multiple Myeloma; Stage III Multiple Myeloma; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia; Untreated Childhood Acute Lymphoblastic Leukemia; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myeloproliferative Syndrome, Transient; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Blastic Plasmacytoid Dendritic Cell Neoplasm; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myelomonocytic, Chronic; Intraocular Lymphoma; Leukemia, Myelomonocytic, Juvenile; Leukemia, Mast-Cell; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Immunoglobulin Light-chain Amyloidosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Multiple Myeloma; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — fludarabine phosphate; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Cyclosporine; Mycophenolic Acid

ARMS (2):
- Arm I (indolent disease) (Experimental): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: Patients undergo donor PBSCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO BID or IV every 8-12 hours on days -3 to 56 with a taper to day 180 and mycophenolate mofetil PO BID or IV every 8-12 hours on days 0 to 27.
  Interventions: Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: peripheral blood stem cell transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis
- Arm II (aggressive disease) (Experimental): CONDITIONING REGIMEN: Patients receive fludarabine phosphate and undergo TBI as in Arm I.
  TRANSPLANTATION: Patients undergo donor PBSCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO BID or IV every 8-12 hours on days -3 to 56 with a taper to day 70 and mycophenolate mofetil as in Arm I.
  Interventions: Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: peripheral blood stem cell transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Procedure: peripheral blood stem cell transplantation — Undergo PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo PBSCT
Drug: cyclosporine — Given PO or IV
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies fludarabine phosphate and total-body radiation followed by donor peripheral blood stem cell transplant and immunosuppression in treating patients with hematologic malignancies. Giving chemotherapy and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving total-body irradiation together with fludarabine phosphate, cyclosporine, and mycophenolate mofetil before transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the rate of grade III/IV graft-versus-host disease (GVHD) in patients treated with low-dose total body irradiation (TBI), fludarabine (fludarabine phosphate), PBSC infusion and immunosuppression with mycophenolate mofetil and a disease risk-based cyclosporine taper.

II. To estimate the risk of graft rejection, GVHD, disease response, non-relapse mortality and the incidence and severity of infectious complications using this treatment strategy.

OUTLINE: Patients are assigned to 1 of 2 treatment groups.

ARM I (indolent disease):

CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) on days -4 to -2 and undergo TBI on day 0.

TRANSPLANTATION: Patients undergo donor peripheral blood stem cell transplantation (PBSCT) on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) twice daily (BID) or IV every 8-12 hours on days -3 to 56 with a taper to day 180 and mycophenolate mofetil PO BID or IV every 8-12 hours on days 0 to 27.

ARM II (aggressive disease):

CONDITIONING REGIMEN: Patients receive fludarabine phosphate and undergo TBI as in Arm I.

TRANSPLANTATION: Patients undergo donor PBSCT on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine PO BID or IV every 8-12 hours on days -3 to 56 with a taper to day 70 and mycophenolate mofetil as in Arm I.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-Hodgkin lymphoma (NHL), chronic lymphocytic leukemia (CLL) or multiple myeloma who are not eligible for a curative autologous transplantation or who have received a prior autologous transplantation; patients with NHL or CLL must have failed prior therapy with an alkylating agent and/or fludarabine, or be at high risk of relapse; patients with multiple myeloma must have stage II or III disease and received prior chemotherapy
* Patients < 50 years of age with NHL, Hodgkin's disease (HD), CLL or multiple myeloma at high risk of regimen related toxicity through prior autologous transplant or through pre-existing medical conditions
* Patients < 75 years of age with other malignant diseases treatable by allogeneic bone marrow transplant (BMT) whom through pre-existing chronic disease affecting kidneys, liver, lungs, and heart are considered to be at high risk for regimen related toxicity using standard high dose regimens; the following diseases are the likely candidates

  * Myelodysplastic syndromes
  * Myeloproliferative syndromes
  * Acute Leukemia with < 10% blasts
  * Amyloidosis
  * Hodgkin's disease
* The Fred Hutchinson Cancer Research Center (FHCRC) Patient Care Conference (PCC) may approve patients with other malignancies or patients declining standard allografts for transplant following presentation and approval; centers outside the FHCRC that have a PCC or equivalent should obtain their Institutional approval; if there is not a comparable group at the Institution, please contact the FHCRC Principal Investigator for FHCRC approval through PCC
* DONOR: Human leukocyte antigen (HLA) genotypically or phenotypically identical related donor
* DONOR: Donor must consent to filgrastim (G-CSF) administration and leukapheresis
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian)

Exclusion Criteria:

* Eligible for a high-priority curative autologous transplant
* Patients with rapidly progressive aggressive NHL unless in minimal disease state
* Any current central nervous system (CNS) involvement with disease
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant
* Patients who are human immunodeficiency virus (HIV) positive
* Cardiac ejection fraction < 40%; ejection fraction is required if the patient has a history of anthracyclines or history of cardiac disease
* Receiving supplementary continuous oxygen
* Diffusing capacity of the lung for carbon monoxide (DLCO) < 30%
* Total lung capacity (TLC) < 30%
* Forced expiratory volume in one second (FEV1) < 30%
* Total bilirubin > 2x the upper limit of normal
* Serum glutamate pyruvate transaminase (SGPT) and serum glutamic oxaloacetic transaminase (SGOT) 4x the upper limit of normal
* Karnofsky score < 50
* Patients with poorly controlled hypertension who are unable to have blood pressure kept below 150/90 on standard medication
* Patients with renal failure are eligible, however patients with renal compromise (serum creatinine greater than 2.0) will likely have further compromise in renal function and may require hemodialysis (which may be permanent) due to the need to maintain adequate serum cyclosporine levels
* The addition of cytotoxic agents for "cytoreduction" with the exception of hydroxyurea and imatinib mesylate will not be allowed within two weeks of the initiation of conditioning
* DONOR: Identical twin
* DONOR: Age less than 12 years
* DONOR: Pregnancy
* DONOR: Infection with HIV
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to G-CSF
* DONOR: Current serious systemic illness

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2000-12; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Probability of severe (grade III/IV) GVHD in each arm | Up to day 84
  95% confidence interval will be calculated.
Probability of severe (grade III/IV) GVHD in each arm | Up to 5 years
  95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
Incidence of graft rejection | Day 28
  Chimerism analysis by fluorescent in situ hybridization (FISH) or variable number tandem repeat (VNTR). Examined and reported in a descriptive manner. Confidence intervals will be presented.
Incidence of graft rejection | Day 56
  Chimerism analysis by FISH or VNTR. Examined and reported in a descriptive manner. Confidence intervals will be presented.
Incidence of graft rejection | Day 84
  Chimerism analysis by FISH or VNTR. Examined and reported in a descriptive manner. Confidence intervals will be presented.
Incidence of graft rejection | Day 180
  Chimerism analysis by FISH or VNTR. Examined and reported in a descriptive manner. Confidence intervals will be presented.
Incidence of graft rejection | Day 365
  Chimerism analysis by FISH or VNTR. Examined and reported in a descriptive manner. Confidence intervals will be presented.
Incidence of non-relapse mortality | Up to 5 years
  Examined and reported in a descriptive manner. Confidence intervals will be presented.
Incidence of infectious complications | Up to 5 years
  Examined and reported in a descriptive manner. Confidence intervals will be presented.
Severity of infectious complications | Up to 5 years
  Examined and reported in a descriptive manner. Confidence intervals will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (11):
- United States (9):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - City of Hope Medical Center, Duarte, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Baylor University Medical Center, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Froedtert Hospital, Milwaukee, Wisconsin
- Universitaet Leipzig, Leipzig, Germany
- University of Torino, Torino, Italy

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241